CLINICAL TRIAL: NCT00446836
Title: Phase II Study of Xyotax in Advanced Hormone Refractory Prostate Cancer
Brief Title: Efficacy and Safety Study of Xyotax to Treat Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Collaborators: Cellular Therapeutics (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PAC IRB#03-0192-05; PCa-X-02 (Other: Principal Investigator)
Record Dates: First submitted 2007-03-12; First posted 2007-03-13 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Prostatic Neoplasms
Keywords: Adenocarcinoma of the prostate; Recurrent prostate cancer; Hormone refractory prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — paclitaxel poliglumex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm (Other): Open label use of Xyotax
  Interventions: Drug: Paclitaxel polyglumex (Xyotax)

INTERVENTIONS:
Drug: Paclitaxel polyglumex (Xyotax) — biologically enhanced chemotherapeutic
  Other Names: Xyotax

SUMMARY:
The purpose of this study is to determine whether Xyotax, a conjugate of the taxane drug paclitaxel, is effective in the treatment of prostate cancer that is no longer responsive to hormone therapy.

DETAILED DESCRIPTION:
Prostate cancer is the second leading cause of cancer death in American men. Hormonal ablation, in the form of medical or surgical castration, is the cornerstone of management for metastatic prostate cancer; however, treatment options for a patient in whom androgen ablation fails are limited. Docetaxel and paclitaxel, taxanes that are cell cycle specific, play a major role in advanced hormone-refractory prostate cancer treatment. In preclinical studies, Xyotax, a conjugate of paclitaxel with enhanced permeability and retention in tumor tissue, has an improved therapeutic profile, with both decreased systemic drug-related toxicities and enhanced efficacy. Xyotax as a single agent has been studied in a broad variety of syngeneic and xenogeneic tumor models. Recognizing that taxanes are active in prostate cancer and preclinical data reports activity with Xyotax in docetaxel and paclitaxel resistant cell lines, there is significant rationale to develop this agent in prostate cancer. Thus, a phase II study is needed to evaluate the antitumor activity in two subsets of hormone refractory prostate cancer patients: those with no prior systemic and those with one prior systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Progressing adenocarcinoma of the prostate having failed prior hormone therapy
* Free of serious co-morbidity
* Have a life expectancy of ≥ 24 weeks
* Maintaining castrate status (either surgically or hormonally)

Exclusion Criteria:

* Patients with central nervous system metastases, except those patients who have had excision or radiotherapy and remain asymptomatic, off steroids and with no evidence of disease as shown by MRI for at least 6 months
* Patients known to be HIV positive
* Patients with active autoimmune disease
* Patients involving concurrent anticancer drug therapy
* Patients with unstable medical condition, such as uncontrolled diabetes mellitus or hypertension; active infections requiring systemic antibiotics, antivirals, or antifungals; clinical evidence of cardiac or pulmonary dysfunction including, but not limited to: unstable CHF, uncontrolled arrhythmias, unstable coagulation disorders, or recent myocardial infarction (within 6 months)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2005-03; Primary Completion 2007-11 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
PSA response | during trial (data from study not available)
  data from study not available
Correlation with soft tissue response | during trial (data from study not available)
  data from study not available

SECONDARY OUTCOMES:
Time to progression | during trial (data from study not available)
  data from study not available

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Amato, DO, Principal Investigator — Baylor College of Medicine - Methodist Hospital
Locations (1):
- Baylor College of Medicine -Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No